CLINICAL TRIAL: NCT05366686
Title: The Effect of NICE Support Program on Frailty and Quality of Life in Patients With Heart Failure
Acronym: NICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ai-Fu Chiou (Other)
Responsible Party: Sponsor-Investigator, Ai-Fu Chiou, Professor, National Yang Ming Chiao Tung University
Organization: National Yang Ming Chiao Tung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YM108131E
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-05

CONDITIONS: Frailty; Quality of Life
Keywords: Frailty; Quality of Life; Heart failure; Exercise program; nutrition
MeSH Terms: conditions — Frailty; Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients in the intervention group will receive a 12 week exercise program including: individual consultation, nutrition consultation, teaching exercise which contain walking and resistance exercise by using elastic bands and elastic balls.
Who Masked: Outcomes Assessor
Masking Description: One research assistant is trained for being a outcomes assessor in this study who did not know the allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frailty and Quality of Life in Patients With Heart Failure (Experimental): Patients in this group will receive a 12 week exercise program including: (1) one 40-60 minute individual consultation (teaching exercise which contain walking and resistance exercise by using elastic bands and elastic balls); (2) provided exercise booklet, exercise log, exercise video; (3) Nutritional consultation; (4) telephone follow-up once per week for 12 weeks
  Interventions: Behavioral: NICE Support Program
- Frailty and Quality of Life (No Intervention): Patients in this group maintain their daily life activities, and there is no intervention given.

INTERVENTIONS:
Behavioral: NICE Support Program — Patients in experimental group will receive a 12 week NICE Support program; patients in control group maintain their usual life activities.
  Arms: Frailty and Quality of Life in Patients With Heart Failure

SUMMARY:
This RCT study aims to examine effects of a NICE Support Program in heart failure patients.

The following hypotheses were tested: patients who received the NICE program will report significant improvement in frailty , social support, anxiety, and depression, quality of life, and nutritional assessment at baseline,4 weeks, 12 weeks and 24 weeks.

DETAILED DESCRIPTION:
This study aims to develop NICE Support program, and examine the effects of an NICE program in heart failure patients. An experimental design is used. Subjects are selected using a purposeful sampling and are randomly assigned to the intervention or control group by using block size randomization method. Patients in the intervention group will receive a 12 week NICE Support program including: individual consultation, nutritional consultation, teaching exercise which contain walking and resistance exercise by using elastic bands and elastic balls. Data are collected by physical indicators and a structural questionnaire to measure frailty, quality of life, social support, anxiety and depression, symptom distress at baseline, 4 weeks, 12 weeks and 24 weeks . Data analysis includes descriptive statistics, Pearson correlation coefficient, independent t test, chi square, one way ANOVA and generalized estimating equation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged above 20 and stable condition and had received physical activity.
2. Clear consciousness, can communicate with Chinese and Taiwanese.
3. Consent to join in this study.
4. Have a smartphone and be able to join social media(Line: heart together-go go go )

Exclusion Criteria:

1. Bed-ridden or unable to perform activities of daily living independently.
2. Unstable illness condition.
3. Emergency condition.
4. Contraindications of performing exercise such as uncontrolled hypertension, uncontrolled arrhythmia.
5. Patients with increased nerve, muscle, bone or rheumatoid diseases due to exercise

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Change Frailty Assessment Scale for Heart Failure, FAS-HF) and Clinical Frailty Scale scores | baseline, 4week, 12 week, 24week
  Changes from baseline Frailty Assessment Scale for Heart Failure, FAS-HF) scores including three indicators: physical, Psychological and social , at 6 weeks, 12 weeks, 24 weeks. FAS-HF scale contains 15 items, each item use Likert scale five point scoring, the total scores ranged from 0 to 45, the higher scores indicate higher frailty.
  Changes from baseline Clinical Frailty Scale including nine indicators, the higher scores indicate higher frailty.
Changes in symptoms distress scores | baseline, 4week, 12 week, 24week
  Changes from baseline symptoms distress scale at 4 weeks, 12 weeks, 24 weeks. Symptoms distress scale contains 17 common symptoms items, each item use Likert scale five point scoring, the total scores ranged from 17 to 85, the higher scores indicate worse symptom distress.

SECONDARY OUTCOMES:
The Minnesota living with heart failure questionnaire(MLHFQ) | baseline, 4week, 12 week, 24week
  Changes from baseline Minnesota living with heart failure questionnaire at 4 weeks, 12 weeks, 24 weeks. The Minnesota living with heart failure questionnaire contains 21 questions regarding the effects of heart failure on patients' physical (eight questions),emotional (five questions) and general (eight questions) dimensions. The possible answer for each question ranges from 0(no) to 5(a lot), and the total score range is 0-105; a higher score indicates lower quality of life .
Changes in anxiety and depression scores | baseline, 4week, 12 week, 24week
  Changes from baseline hospital anxiety and depression scale at 6 weeks, 12 weeks, 24 weeks. The hospital anxiety and depression scale contains 14 questions(7 for assess anxiety and 7 for assess depression), each item use Likert scale four point scoring, the total scores ranged from 0 to 21, the higher scores indicate more severe anxiety and depression level.

CONTACTS AND LOCATIONS:
Overall Officials: Ai-Fu Chiou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afilalo, J. (2019). Evaluating and treating frailty in cardiac rehabilitation. Clinics in Geriatric Medicine, 35(4), 445-457. https://doi.org/10.1016/j.cger.2019.07.002. PMID: 31543177 Afilalo J, Alexander KP, Mack MJ, Maurer MS, Green P, Allen LA, Popma JJ, Ferrucci L, Forman DE. (2014). Frailty assessment in the cardiovascular care of older adults. Journal of the American College of Cardiology, 63(8), 747-762. https://doi.org/10.1016/j.jacc.2013.09.070. PMID: 24291279 Denfeld QE, Winters-Stone K, Mudd JO, Gelow JM, Kurdi S, Lee CS. (2017). The prevalence of frailty in heart failure: A systematic review and meta-analysis. The International Journal of Cardiology, 236, 283-289. PMID: 28215466 Flint KM, Pastva AM, Reeves GR. (2019). Cardiac rehabilitation in older adults with heart failure: Fitting a square peg in a round hole. Clinics in Geriatric Medicine, 35(4), 517-526. https://doi.org/10.1016/j.cger.2019.07.008. PMID: 31543182
- [Derived] Wang TC, Hsieh YC, Yang CY, Lee CM, Liu CY, Chiou AF. Effects of a multimodal support intervention (the NICE-Support programme) on frailty and quality of life in patients with heart failure: a randomized controlled trial. Eur J Cardiovasc Nurs. 2026 Jan 3:zvaf187. doi: 10.1093/eurjcn/zvaf187. Online ahead of print. PMID 41482005